CLINICAL TRIAL: NCT03822572
Title: ABCSG C08 - Exercise II: Randomized Trial of Endurance Exercise Following Adjuvant Chemotherapy for Colorectal Cancer
Brief Title: ABCSG C08-Exercise II: Trial of Endurance Exercise Following Adjuvant Chemotherapy for Colorectal Cancer
Acronym: ABCSG C08
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Oberösterreichische Krebshilfe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ABCSG C08
Record Dates: First submitted 2018-11-29; First posted 2019-01-30 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Carcinoma
Keywords: endurance exercise
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A - endurance exercise (Experimental): All patients receive a pulse-controlled endurance exercise program based on the study results by O'Donovan. The individual pulse-controlled endurance exercise should be performed 3 times a week. On the basis of age, weight, sex and body fat the normal weight will be calculated. The kilocalories (kcal), which correspond to the metabolic equivalent task (MET) hour per week, will be calculated after age and gender adjustment of the normal weight. The endurance exercise will be increased gradually until reaching 18 MET-hours/wk during the year of endurance exercise. Patients in arm A can perform different types of endurance exercise (bicycling, cross walking, jogging, walking, nordic walking, cross country skiing)
  Interventions: Other: endurance exercise
- B - control arm (Other): Patients in this arm should maintain their habitual physical activity pattern as before the diagnoses of colorectal cancer.
  Interventions: Other: control

INTERVENTIONS:
Other: endurance exercise — defined exercise program
  Arms: A - endurance exercise
Other: control — habitual physical activity before the diagnosis
  Arms: B - control arm

SUMMARY:
ABCSG C08 is a randomized, two-arm, multicenter trial to investigate the efficacy of endurance exercise following adjuvant chemotherapy in patients with colorectal cancer.

Indication: Locally advanced colorectal cancer after adjuvant chemotherapy. Evidence supporting the beneficial effects of exercise programs during chemotherapy are available, the results across studies are not entirely consistent. Additional studies are needed to determine the optimal content, intensity, and form of training programs.

DETAILED DESCRIPTION:
Colorectal cancer is the second leading cause of cancer mortality in Western countries after breast cancer among women and lung cancer among men. About 5.000 new cases are diagnosed each year in Austria. This represents an annual incidence of 50-60 per 100.000 inhabitants. In patients with colorectal cancer stage III and in certain situations even in stage II adjuvant chemotherapy is indicated after R0 resection. Despite recent advances in adjuvant chemotherapy 20-30% of these patients still relapse. About 80% of recurrences occur in the first three years.

There is consistent evidence from several observational epidemiologic studies that physical activity reduces the risk of developing colon cancer. In recent years several observational studies even showed a reduction in relapse rate, colon cancer-specific mortality and overall mortality by physical activity in patients with colon and breast cancer. Colon cancer survivors who engaged in higher levels of physical activity experienced a 50-60% improvement in long-term outcomes compared to inactive patients. Different mechanisms for the protective effect of physical activity on colon cancer have been proposed and it is believed that the same mechanisms of physical activity are also involved in the improvement of disease outcomes in gastrointestinal cancer survivors. Physical activity leads to decrease of inflammation, decreased levels of insulin-like growth factor (IGF) and insulin, reduced transit time through the gut and increased levels of vitamin D. Factors, that are associated with a reduced risk of colon polyps, colon cancer and colon cancer mortality.

A review on the impact of various exercise programs on fatigue, found good evidence that exercise not only decreased levels of fatigue, but also increased quality of life, mood and functioning.

While there is evidence supporting the beneficial effects of exercise programs during chemotherapy, the results across studies are not entirely consistent. Additional studies are needed to determine the optimal content, intensity, and form of training programs.

Recently ABCSG has investigated the feasibility of endurance exercise after adjuvant chemotherapy in patients with locally advanced colorectal cancer in the investigator's study group (ABCSG C07 Exercise - pilot study). Results concerning compliance of patients have been considered for sample size estimations and study planning.

ELIGIBILITY:
Inclusion Criteria:

* completely resected, histologically confirmed adenocarcinoma of the colon or rectum
* patients, who have completed adjuvant chemotherapy 4-16 weeks prior to randomization
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Age ≥18 years
* adequate hematologic functions <=28d prior to randomization
* able to perform endurance exercise according to protocol
* ability to perform ergometry in order to assess physical capability at the discretion of the investigator
* signed informed consent prior to randomization

Exclusion Criteria:

* significant comorbid conditions precluding participation in a physical activity program (investigators decision)
* disabled patients unable to participate in the physical activity program
* Regular (3-times a week) vigorous physical activity of >150 minutes (type of physical activity: bicycling, cross walking (cross trainer), jogging, walking at a brisk pace, nordic walking, cross country skiing) within the last year before diagnosis of colorectal cancer
* patients unwilling to complete endurance exercise or complete all questionnaires related to the study
* past or current history of other malignant neoplasms other than colorectal cancer in the last 5 years except basal cell carcinoma of the skin and/or in situ carcinoma of the cervix
* clinically significant cardiovascular disease
* left bundle branch block
* current study with chemotherapy or radiation
* current pregnancy or plans to become pregnant within the next 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint - disease free survival (DFS) | 8 years (after Last Patient Out (LPO))
  DFS is defined as the time from randomization to locoregional or metastatic recurrence or the appearance of secondary cancer or death, whichever occurs first. Recurrence may be either histologically proven or evidenced by imaging via MRI or CT. Isolated CEA evaluation will not be sufficient to determine a relapse.

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint I - relapse free survival (RFS) | 8 years (after Last Patient Out (LPO))
  RFS is defined as the time from randomization to locoregional or metastatic recurrence of colorectal cancer or death, whichever occurs first
Secondary Efficacy Endpoint II - overall survival (OS) | 8 years (after Last Patient Out (LPO))
  OS is defined as time from randomization to death from any cause
Physical Activity Endpoint I - physical activity measured by MET-hours | 8 years (after Last Patient Out (LPO))
  Evaluation of physical activities measured by MET-hours in the domains "work", "leisure time ", "sedentary behavior" and "transporation" by Global Physical Activity Questionnaire (GPAQ) within each study arm and compared between study arms at baseline, at 3, at 6, at 12, at 24 and at 36 months
Physical Activity Endpoint II - endurance exercise measured by MET-hours | 8 years (after Last Patient Out (LPO))
  Evaluation of endurance exercise measured by MET-hours by pulse-control in arm A at 3, at 6 and at 12 months
Physical Activity Endpoint III - performance enhancement measured by MET-hours by ergometry | 8 years (after Last Patient Out (LPO))
  Evaluation of performance enhancement measured by MET-hours by ergometry within each study arm (arm A at baseline, at 3, at 6 and at 12 months; arm B at baseline and at 12 months) and compared between study arms at baseline and at 12 months
Physical Activity Endpoint IV - physical activity measures | 8 years (after Last Patient Out (LPO))
  Correlation of MET-hours in the domains "work", "leisure time ", "sedentary behavior" and "transporation" by Global Physical Activity Questionnaire (GPAQ) and results of endurance exercise as well as performance enhancement by ergometry (both measured by MET-hours) with DFS, RFS and OS
Patient Reported Outcome Endpoint I - fatigue | 8 years (after Last Patient Out (LPO))
  Evaluation of fatigue as measured by EORTC - QLQ FATIGUE CAT Theta scores compared between study arms. Score has no fixed upper and lower limit and a high score represents a high level of fatigue.
Patient Reported Outcome Endpoint II - emotional functioning score | 8 years (after Last Patient Out (LPO))
  Evaluation of the emotional functioning score (based in the functional scale EF) as measured by EORTC QLQ-C30 emotional functioning (based on items) compared between study arms, where a high score for a functional scale represents a high/healthy level of functioning.
Patient Reported Outcome Endpoint III - physical functioning score | 8 years (after Last Patient Out (LPO))
  Evaluation of the standardized physical functioning score (based on the revised functional scale PF2) as measured by EORTC QLQ-C30 physical functioning compared between study arms, where a high score for a functional scale represents a high/healthy level of functioning
Patient Reported Outcome Endpoint IV - global quality of life (QoL) score | 8 years (after Last Patient Out (LPO))
  Evaluation of the standardized global health status/QoL score (based on the revised global health status/QoL QL2) as measured by EORTC QLQ-C30 summary score compared between study arms, where a high score for the global health status/QoL represents a high QoL.
Patient Reported Outcome Endpoint V - patient reported outcomes (fatigue, emotional functioning, physical functioning, global quality of life) | 8 years (after Last Patient Out (LPO))
  Correlation of all patient reported outcomes explained above (fatigue, emotional functioning, physical functioning, global quality of life) with MET-hours
Body Composition Endpoint I - body mass index (BMI) | 8 years (after Last Patient Out (LPO))
  Evaluation of the influence of BMI on DFS, RFS and OS
Body Composition Endpoint II - body fat | 8 years (after Last Patient Out (LPO))
  Evaluation of the influence of body fat on DFS, RFS and OS
Body Composition Endpoint III - waist circumference | 8 years (after Last Patient Out (LPO))
  Evaluation of the influence of waist circumference on DFS, RFS and OS
Cardiovascular Endpoint - cardiovascular complications | 8 years (after Last Patient Out (LPO))
  Evaluation of the incidence of cardiovascular complications (myocardial infarction, stroke, newly diagnosed diabetes mellitus, newly diagnosed hypertension)
Safety Endpoint I - serious adverse events (SAEs) | 8 years (after Last Patient Out (LPO))
  Evaluation of the incidence of physical activity related SAEs and physical activity related deaths in both arms
Safety Endpoint II - time to SAEs | 8 years (after Last Patient Out (LPO))
  Evaluation of time from study start to physical activity related SAEs
Exploratory Endpoint - molecular and biochemical markers (will be defined during the course of the study) | 8 years (after Last Patient Out (LPO))
  Correlation of molecular and biochemical markers with DFS, RFS, OS and with physical activity. The analysis of molecular markers will depend on the markers which will be defined during the course of the study in addition to Insulin & ILGF.

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Piringer, MD, MSc, Study Chair — Austrian Breast & Colorectal Cancer Study Group
Locations (8):
- Austria (8):
  - LKH Salzburg-PMU, UNiv. KLinik f. Innere Med III, Salzburg, Salzburg
  - Med. Univ. Graz, Graz, Styria
  - BKH Kufstein, Kufstein, Tyrol
  - KH St. Josef Braunau, Braunau am Inn, Upper Austria
  - Hospital BHS Linz, Coop. Study Group, Linz, Upper Austria
  - Kepler Universitätsklinikum Linz, Linz, Upper Austria
  - Pyhrn-Eisenwurzen Klinikum Steyr, Steyr, Upper Austria
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria

IPD SHARING:
Plan to Share IPD: No
currently sharing of IPDs (Individual Participant Data) is not planned in this trial